CLINICAL TRIAL: NCT04386993
Title: De-escalated Conformal Radiation Expedited Sequentially With Chemotherapy for Endometrial Cancer (DeCRESCEndo)
Brief Title: De-escalated Conformal Radiation Expedited Sequentially With Chemotherapy for Endometrial Cancer
Acronym: DeCRESCEndo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202004237
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- IMRT (Experimental): -Five 5-Gy fractions of IMRT will be given to the pelvis with elective simultaneous boost to any suspicious lymph node or residual disease to 30 Gy.
  -*Brachytherapy boost (at the discretion of the PI) within 2 weeks of radiation therapy completion. Once or twice weekly for three weeks
  Interventions: Radiation: Intensity modulated radiation therapy

INTERVENTIONS:
Radiation: Intensity modulated radiation therapy — Radiation should be delivered over the course of 1-2 weeks (allowing for weekends/holidays).
  Other Names: IMRT

SUMMARY:
The goal of this study is to evaluate short course radiation in the post-operative female pelvis after hysterectomy in stage III-IVA endometrial adenocarcinoma patients, or any stage patients with uterine serous or carcinosarcoma histology. The investigators hypothesize that short course pelvic radiation will have an acute and late grade 3-4 toxicity rate < 10%, and patients will benefit from both convenient and effective loco-regional control comparable to the traditional 5-6 weeks of radiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IIIA-IVA endometrial cancer, or any stage I-IVA where any proportion of the tumor is uterine serous, clear cell, de-differentiated, or carcinosarcoma histology.
* Must have already undergone radical hysterectomy. Hysterectomy may have occurred no more than one year prior to enrollment.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Minimal bone marrow and organ function as defined below:

  * Leukocytes ≥ 1,000 cumm
  * Absolute neutrophil count ≥ 500 cumm
  * Platelets ≥ 50,000 cumm
  * Hemoglobin ≥ 7g/dL
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior radiation to the pelvis.
* Currently receiving any investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, inflammatory bowel disease, or irritable bowel disease.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Incidence of acute hematologic, gastrointestinal, and genitourinary adverse events | From start of radiation through Day 90
Incidence of late hematologic, gastrointestinal, and genitourinary adverse events | From Day 91 through month 12

SECONDARY OUTCOMES:
Change in patient-reported urinary and gastrointestinal toxicity as measured by PRO-CTCAE | Baseline, 2 weeks, and 3 months post-completion of radiation
  * PRO-CTCAE responses are scored from 0 to 4 with 0=Never/Not at all/None and 4=Frequently/Very Much/Very Severe/Almost Constantly
  * Scores for each attribute (frequency, severity and/or interference) will be presented descriptively
Change in patient-reported urinary and gastrointestinal toxicity as measured by bowel/bladder domains of EPIC-26 | Baseline, 2 weeks, 3 months, 6 months, and 12 months post-completion of radiation
  * Bladder has 7 questions and bowel has 9 questions
  * The response for each item is standardized to a 0 to 100 scale
  * The standardized values will be averaged for all items within a group to create the summary or subscale score.
Change in quality of life as measured by FACT-En | Baseline, 2 weeks, 3 months, 6 months, and 12 months post-completion of radiation
  * Questionnaire asking questions about physical well-being, social/family well-being, emotional well-being, functional well-being, and other additional concerns. Answers range from 0 = not at all to 4 = very much. Questions are phrased so that higher numbers indicate a better health state,
  * Scoring is performed through a simple sum of item scores. Each subscale is scored, and a total score is obtained by adding each of the subscale scores.
Locoregional control | Up to 12 months post-completion of radiation
  -Locoregional recurrence is defined as histologic or radiographic evidence of cancer in the previously resected site or regional lymph nodes included in the radiated field.
Distant control | Up to 12 months post-completion of radiation
  -Distant recurrence is defined as histologic or radiographic evidence of cancer outside of the radiated field.
Disease-free survival | Up to 12 months post-completion of radiation
  -Disease-free survival is defined as survival with no evidence of disease recurrence or death
Overall survival | Up to 12 months post-completion of radiation
  -Number of participants alive at the time of completion of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jessika Contreras, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices) for individual participant data meta-analysis by investigators whose proposed use of data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
Supporting Information: Study Protocol
Time Frame: Proposals may be submitted up to 36 months following article publication.
Access Criteria: Please contact Dr. Jessika Contreras.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu